CLINICAL TRIAL: NCT05438264
Title: Effect of Donepezil on Speech Recognition in Cochlear Implant Users
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Aaron Moberly, Professor, Otolaryngology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 220844
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Bilateral Sensorineural Hearing Loss
Keywords: cochlear implant; sensorineural hearing loss; donepezil
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Donepezil 5 mg, daily
  Interventions: Drug: Donepezil
- Control (Placebo Comparator): Placebo, daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil — acetylcholinesterase inhibitor
  Other Names: Aricept
  Arms: Experimental
Drug: Placebo — placebo
  Arms: Control

SUMMARY:
Hearing loss is a major cause of disability that affects over 48 million Americans. There are currently no medications used to treat sensorineural hearing loss. Cochlear implants can significantly restore hearing in adults with moderate to profound sensorineural hearing loss, but their utility is limited by the wide variability in hearing outcomes. Differences in cochlear implant outcomes may be explained by neuroplasticity, as neural networks must reorganize to process the new auditory information provided by the implant.

The investigators predict that cholinergic enhancement with donepezil (an acetylcholinesterase inhibitor) may facilitate cortical reorganization in cochlear implant users, leading to functional improvements in speech recognition and cognition. In addition to taking donepezil, study participants will be asked to increase their daily processor use. Studies suggest that increasing daily device use can improve speech recognition, and this study will explore whether this effect can be augmented further with donepezil.

In this randomized, double-blind controlled trial, the investigators aim to assess the effects of donepezil on speech recognition, cortical plasticity, and cognition. Participants will start daily treatment with either donepezil 5 mg or placebo. Participants will be followed longitudinally at 1 month and 3 months after starting the study. The findings from this study will provide important insight into the mechanisms of hearing restoration and could potentially improve hearing and cognitive outcomes for future cochlear implant users.

DETAILED DESCRIPTION:
The proposed study is a double-blind, randomized controlled trial comparing donepezil with placebo in adult cochlear implant users.

Aim 1: Evaluate if donepezil treatment improves speech recognition in cochlear implant users.

Aim 2: Evaluate if donepezil treatment increases intramodal auditory cortex activity in cochlear implant users.

Aim 3: Evaluate if donepezil treatment improves cognition in cochlear implant users.

ELIGIBILITY:
Inclusion Criteria:

1. At least 6 months of cochlear implant use
2. Age ≥ 18 years
3. Post-lingual onset of deafness
4. Audiometric thresholds meeting FDA-labeled indications for adult cochlear implantation
5. Normal or corrected-to-normal vision assessed with a Snellen eye chart
6. English verbal communication
7. No participation in any other clinical trial within the past 3 months
8. Physically healthy
9. Female participants must have no child-bearing potential or agree to practice effective contraception during the study (such as established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; condom with spermicidal foam/gel/film/cream/suppository; occlusive cap with spermicidal foam/gel/film/cream/suppository; male partner sterilization; or true abstinence when this is in line with the preferred and usual lifestyle of the subject)
10. Female participants of child-bearing potential must have a negative urine pregnancy test at the time of enrollment and before each study visit

Exclusion Criteria:

1. Evidence of conductive hearing loss
2. Diagnosed neurological or sensory disorder (such as Alzheimer's disease, Parkinson's disease, epilepsy, stroke, autism, schizophrenia, or uncorrected visual impairment)
3. Positive urine pregnancy test at any time during the study
4. Breastfeeding or nursing at any time during the study
5. Known hypersensitivity to donepezil hydrochloride or to piperidine derivatives
6. Current use of medications with known anticholinergic effects (such as tricyclic antidepressants, first-generation antihistamines, or bladder antispasmodics)
7. Current or prior use of cholinesterase inhibitors
8. Use of tobacco or nicotine products in the past 1 month
9. Severe anatomic abnormalities of the temporal bone
10. Major active life-threatening illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative monosyllabic word recognition | 3 months
  Monosyllabic word recognition using consonant-nucleus-consonant (CNC) word lists

SECONDARY OUTCOMES:
Cognitive outcome | 3 months
  NIH Cognitive Toolbox and Repeatable Battery for the Assessment of Neuropsychological Status for Hearing Impaired Individuals

CONTACTS AND LOCATIONS:
Overall Officials: René Gifford, PhD, Principal Investigator — Vanderbilt University Medical Center; Mark Wallace, PhD, Principal Investigator — Vanderbilt University; Aaron Moberly, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will share raw de-identified summary data upon request.